CLINICAL TRIAL: NCT03590067
Title: Oral Findings in a Group of Egyptian Pediatric Patients at Endstage Renal Disease Either on Haemodialysis or After Renal Transplantation
Brief Title: Oral Findings in a Group of Egyptian Pediatric Patients at Endstage Renal Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rahma Ali Saber Ali, Dentist, Cairo University
Other Study IDs: CEBD-CU-2018-06-26
Record Dates: First submitted 2018-06-29; First posted 2018-07-18 (Actual); Last update posted 2019-07-31 (Actual); Status verified 2019-07

CONDITIONS: Kidney Disease, Chronic
Keywords: End stage renal disease; Haemodialysis; Renal transplantation; pediatric; chronic kidney disease; oral finding; oral manifestation
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic; Oral Manifestations | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heamodialysis group
  Interventions: Other: Questionnaire
- Kidney transplantation group
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The data will be collected through a questionnaire that will be obtained through an interview between the investigator and the parent or the legal guardian

SUMMARY:
In Egypt, the prevalence of end stage renal disease in pediatric population has never been estimated on a national scale. The patients at end stage renal disease encounter oral and dental problems that emphasize regular and careful screening . In Egypt, the prevalence of oral findings is not studied so we conduct this study to study the oral findings among a group of pediatric patients at end stage renal disease either on haemodialysis or after kidney transplantation.

DETAILED DESCRIPTION:
Study setting:

* The study will be held at the center of Pediatric Nephrology and transplantation, El- Mounira children's hospital (Abu El rish).
* The data collected through the questionnaire will be obtained through an interview between the investigator and the parent or the legal guardian that's based on WHO guide for health surveys(WHO Oral health surveys, 2013)
* For patients undergoing dialysis, examination will be performed at the dialysis unit during dialysis session (there is no waiting room for patients before dialysis).
* For patients who received renal transplantation, examination will be performed at the outpatient nephrology clinic during follow up visits.
* Clinical examination will be performed for both oral (soft tissue) and dental (hard) tissue.
* Decayed-Missing-Filled Index ( DMF ) which was introduced by Klein, Palmer and Knutson in 1938 and modified by WHO.

The components are:

D component:

Used to describe (Decayed teeth) which include:

Carious tooth. Filled tooth with recurrent decay. Only the roots are left. Defect filling with caries. Temporary filling. Filled tooth surface with other surface decayed.

M component:

Used to describe (Missing teeth due to caries) other cases should be excluded.

F component:

Used to describe (Filled teeth due to caries). Teeth were considered filled without decay when one or more permanent restorations were present and there was no secondary (recurrent) caries or other area of the tooth with primary caries. A tooth with a crown placed because of previous decay was recorded in this category. Teeth stored for reason other than dental caries should be excluded.

deft / defs , which was introduced by Gruebbel in 1944

d- decayed tooth . e- decayed tooth indicated for extraction . f- filled tooth

• The coding system for the Modified DDE Index has three items of information that will be recorded for each tooth surface. (Clarkson and O'Mullane, 1989)

First, the Type of Defect, codes 0-7, was recorded. Then the Sub-type of that defect was noted, i.e., when a demarcated opacity was present, the Sub-type was either white/cream (code 1) or yellow/brown (code 2), or when a diffuse opacity was present, then six options were possible. Finally, the extent of each defect was recorded. The new additional sub-type (code 3) termed "diffuse confluent opacity" is defined as a diffuse opacity in which any patchiness has merged into a regular condensed chalky white area, and it could cover the entire surface of a tooth or be confined to a localized area of the tooth surface.

* Oral candidiasis assessment will be based on the Lehner scale (Cleverson et al., 2014)
* In assessing the degree of gingival hyperplasia we will use the index of Angelopoulos and Goaz, described by Prof. T. Djemileva. (Dencheva et al., 2011)

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric patients <15 years old with a diagnosis of end stage renal disease "stage 5" receiving dialysis.
2. Pediatric Patients < 15 years old with kidney transplantation in the monthly follow up.
3. Recorded data for every patient. (Glomerular Filtration Rate, Creatinine level, urea level and calcium level).

Exclusion Criteria:

1. Patients undergoing renal dialysis for reasons other than chronic kidney disease, such as acute renal failure secondary to accidents, trauma, snake poisoning.
2. Patients undergoing peritoneal dialysis.
3. Patients not physically able to participate in the examination.
4. Chronic kidney disease patients at stage 2, 3 and 4.

Ages: 2 Years to 14 Years | Sex: All
Age Groups: Child
Study Population: All pediatric patients at end stage renal disease attending at the center of Pediatric Nephrology and transplantation, El- Mounira children's hospital (Abu El rish) will be enrolled in the study in a consecutive order according to inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-01-01 (Estimated)

PRIMARY OUTCOMES:
Caries | Five minutes
  Clinical examination will be done and Caries index will be used ,Unit is the tooth to determine if there is caries or not

SECONDARY OUTCOMES:
Enamel hypoplasia | Ten minutes
  Clinical examination will be done on each patient to assess enamel hypoplasia and recorded by use of Modified Developmental Defect of Enamel (DDE) Index
Oral candidiasis | Five minutes
  Clinical examination will be conducted to assess oral candidiasis and recorded by use of Lehner Oral Candidiasis Classification
Gingival overgrowth | Five minutes
  Clinical examination will be done to asess gingival overgrowth and recorded by use of Angelopoulos and Goaz index

IPD SHARING:
Plan to Share IPD: Undecided